CLINICAL TRIAL: NCT02475187
Title: Observational Study of Thrombogenic Properties in 220 Patients With Proximal Femur Fracture
Acronym: thro-fract15
Status: Terminated | Type: Observational
Sponsor: Vestre Viken Hospital Trust (Other)
Responsible Party: Sponsor
Other Study IDs: REK 2015/139
Record Dates: First submitted 2015-05-31; First posted 2015-06-18 (Estimated); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Thromboembolism
Keywords: TEG; MEA; Thrombotic events; VTE; LMWH; Hip fractures
MeSH Terms: conditions — Thromboembolism; Hip Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood tests for Measurments of thrombotic properies. No storage of specimens
Oversight: Data Monitoring Committee: No

SUMMARY:
Measurement of thrombogenic properties by TEG and MEA and observation of thrombotic events over 2 years in 220 patients with hip fracture.

DETAILED DESCRIPTION:
Patients with proximal femur fracture have high incidences of thrombotic events. By the two "bed-side" methods TEG (Thrombelastography) and MEA (Multiple Electrode Aggregometry), the thrombogenic properties of 220 patients with proximal femur fracture will be measured at time of hospital admission and 4 times over a period of 6 months postoperatively, and the patients will be followed in a total length of 2 years to register thrombotic events.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years who are admitted to our hospital for orthopedic surgery of proximal femur fracture.
* The study participants must be capable to sign/accept informed concent

Exclusion Criteria:

* Patients with severe dementia or that of other causes not ar capable to give informed concent.
* Patients with known or suspected cancer, blood diseases or bleeding disorders
* Surgery last 6 months
* Severe renal- (eGFR (creatinine) <30)
* Severe hepatic failure (2x UNL for bilirubin, 3x UNL for ALAT or INR > 1,3 without anticoagulation treatment)
* Patients that, by drug spesification or -SPC, not are eligible for postoperative thrombosis prophylaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to our hospital for proximal femur fracture and receive orthopedic surgery with concomittant thrombosis prophylaxis with LMWH or anticoagulation with Warfarin, and are capable to sign/accept informed concent
Sampling Method: Non-Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Measurements of thrombogenic properties by TEG (Maximum Amplitude) and MEA (Units) and thrombotic events in 220 patients with Hip Fracture. | 24 months
  Thrombogenic properties measured by TEG (different measurements as "MA") and MEA (measured as "U") 6 months after operation for hip fracture and clinical thrombotic events over 24 months

SECONDARY OUTCOMES:
Measurements of thrombogenic properties by TEG (Maximum Amplitude) and MEA (Units) in 220 patients with Hip Fracture. | 6 months
  Measurements of thrombogenic properties by TEG and MEA in 220 patients patients with Hip Fracture to investigate any correlation between the two Methods and anti-fXa titer.
Measurements of thrombogenic properties by TEG (Maximum amplitude) and MEA (Units)) in the 100 patients with Hip Fracture and thrombotic complications | 6 months
  Measurements of thrombogenic properties by TEG and MEA (in the first) 100 patients with Hip Fracture and .

CONTACTS AND LOCATIONS:
Overall Officials: Øystein Meen, Phd, Principal Investigator — Kongsberg Hospital, Vestre Viken Hospital trust
Locations (1):
- Kongsberg Hospital, Vestre Viken Hospital Trust, Kongsberg, Norway

REFERENCES:
- [Background] Dahl OE, Caprini JA, Colwell CW Jr, Frostick SP, Haas S, Hull RD, Laporte S, Stein PD. Fatal vascular outcomes following major orthopedic surgery. Thromb Haemost. 2005 May;93(5):860-6. doi: 10.1160/TH04-11-0769. PMID 15886800
- [Background] Cattaneo M. Resistance to anti-platelet agents. Thromb Res. 2011 Feb;127 Suppl 3:S61-3. doi: 10.1016/S0049-3848(11)70017-2. PMID 21262444
- [Background] McCrath DJ, Cerboni E, Frumento RJ, Hirsh AL, Bennett-Guerrero E. Thromboelastography maximum amplitude predicts postoperative thrombotic complications including myocardial infarction. Anesth Analg. 2005 Jun;100(6):1576-1583. doi: 10.1213/01.ANE.0000155290.86795.12. PMID 15920177
- [Background] Paniccia R, Antonucci E, Maggini N, Romano E, Gori AM, Marcucci R, Prisco D, Abbate R. Assessment of platelet function on whole blood by multiple electrode aggregometry in high-risk patients with coronary artery disease receiving antiplatelet therapy. Am J Clin Pathol. 2009 Jun;131(6):834-42. doi: 10.1309/AJCPTE3K1SGAPOIZ. PMID 19461090
- [Background] Tantry US, Bonello L, Aradi D, Price MJ, Jeong YH, Angiolillo DJ, Stone GW, Curzen N, Geisler T, Ten Berg J, Kirtane A, Siller-Matula J, Mahla E, Becker RC, Bhatt DL, Waksman R, Rao SV, Alexopoulos D, Marcucci R, Reny JL, Trenk D, Sibbing D, Gurbel PA; Working Group on On-Treatment Platelet Reactivity. Consensus and update on the definition of on-treatment platelet reactivity to adenosine diphosphate associated with ischemia and bleeding. J Am Coll Cardiol. 2013 Dec 17;62(24):2261-73. doi: 10.1016/j.jacc.2013.07.101. Epub 2013 Sep 27. PMID 24076493
- [Background] Sibbing D, Schulz S, Braun S, Morath T, Stegherr J, Mehilli J, Schomig A, von Beckerath N, Kastrati A. Antiplatelet effects of clopidogrel and bleeding in patients undergoing coronary stent placement. J Thromb Haemost. 2010 Feb;8(2):250-6. doi: 10.1111/j.1538-7836.2009.03709.x. Epub 2009 Nov 28. PMID 19943882
- [Background] Kornblith LZ, Kutcher ME, Redick BJ, Calfee CS, Vilardi RF, Cohen MJ. Fibrinogen and platelet contributions to clot formation: implications for trauma resuscitation and thromboprophylaxis. J Trauma Acute Care Surg. 2014 Feb;76(2):255-6; discussion 262-3. doi: 10.1097/TA.0000000000000108. PMID 24458031
- [Background] Wurtz M, Hvas AM, Christensen KH, Rubak P, Kristensen SD, Grove EL. Rapid evaluation of platelet function using the Multiplate(R) Analyzer. Platelets. 2014;25(8):628-33. doi: 10.3109/09537104.2013.849804. Epub 2013 Nov 18. PMID 24246241
- [Background] Wilson D, Cooke EA, McNally MA, Wilson HK, Yeates A, Mollan RA. Changes in coagulability as measured by thrombelastography following surgery for proximal femoral fracture. Injury. 2001 Dec;32(10):765-70. doi: 10.1016/s0020-1383(01)00139-5. PMID 11754883
- [Background] Harr JN, Moore EE, Chin TL, Ghasabyan A, Gonzalez E, Wohlauer MV, Banerjee A, Silliman CC, Sauaia A. Platelets are dominant contributors to hypercoagulability after injury. J Trauma Acute Care Surg. 2013 Mar;74(3):756-62; discussion 762-5. doi: 10.1097/TA.0b013e3182826d7e. PMID 23425732
- [Background] Talsnes O, Hjelmstedt F, Dahl OE, Pripp AH, Reikeras O. Clinical and biochemical prediction of early fatal outcome following hip fracture in the elderly. Int Orthop. 2011 Jun;35(6):903-7. doi: 10.1007/s00264-010-1149-7. Epub 2010 Nov 16. PMID 21079953